CLINICAL TRIAL: NCT04068064
Title: Efficacy and Mechanisms Underlying Emotional Association Bias Modification in Individuals With IGD
Brief Title: Emotional Association Bias Modification Training in Individuals With IGD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Beijing Normal University (Other)
Responsible Party: Principal Investigator, Jin-tao Zhang, Professor, Beijing Normal University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: EABMT_IGD
Record Dates: First submitted 2019-08-20; First posted 2019-08-28 (Actual); Last update posted 2022-07-05 (Actual); Status verified 2022-06

CONDITIONS: Internet Gaming Disorder
MeSH Terms: conditions — Internet Addiction Disorder

STUDY DESIGN:
Intervention Model Description: a randomized, between-subject design, including an intervention group and a control group
Who Masked: Participant, Investigator
Masking Description: the grouping is blind to both participants and the investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- EABM training group (Experimental): about 40 individuals with IGD will be randomly assigned to the EABM training group
  Interventions: Procedure: EABM training
- Control training group (Placebo Comparator): about another 40 individuals with IGD will be randomly assigned to the control training group
  Interventions: Procedure: sham training

INTERVENTIONS:
Procedure: EABM training — The training aims at associating gaming pictures with negative words and pictures of healthy activities with positive words. Gaming pictures are always presented with a pair of negative words. Pictures of healthy activities are always presented with a pair of positive words. Each picture is presented with a fixed pair of words. Participants will be instructed to select one word to get the most monetary reward. Specifically, in response to each gaming picture, selecting one word will have a 70% chance to get a monetary reward and the other word will have a 30% chance to get a monetary reward. A similar rationale applies to the pictures of healthy activities. The reward setting will help consolidate target associations.
  Each training session includes 300 times/trials of each type of association, presented in pseudorandom way. The whole training includes 6 training sessions. Participants will receive one training session every days.
  Arms: EABM training group
Procedure: sham training — In the control group, neutral words instead of emotional words are used. All other settings are the same with those in the intervention group
  Arms: Control training group

SUMMARY:
This project aims to investigate (1) the efficacy of emotional association bias modification (EABM) training on internet gaming disorder (IGD); (2) the underlying neural mechanisms of such efficacy

DETAILED DESCRIPTION:
As with the efficacy, the experiment aims to test whether EABM training will reduce positive emotional association bias towards gaming, compulsive choice of gaming pictures, cue-induced craving for gaming, the severity of gaming behaviors in individuals with IGD.

As with the underlying neural mechanisms, the experiment aims to test whether EABM training will alter the activation of reward circuits in response to gaming pictures, the activation of executive control network (mainly refering to the prefrontal cortex) regarding regulation ability for craving and response inhibition ability.

ELIGIBILITY:
Inclusion Criteria:

1. the 5th edition of Diagnostic and Statistical Manual of Mental Disorders (DSM-5 ) recommended diagnosis of Internet gaming disorder :

   the scores of the 9 items of DSM-5 recommended diagnosis for Internet gaming disorder ≥ 5.

   engagement in popular Internet games (e.g. Arena of Valor, League of Legends and Player Unknown's Battle Grounds) for over 20 hours per week for a minimum of 12 months.
2. the scores of the Young-Internet addiction Test ≥ 50

Exclusion Criteria:

1. current or history of use of illegal substances and other addictions;
2. current or history of psychiatric or neurological illness;
3. current use of psychotropic medications.

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 87 (Actual)
Dates: Start 2019-08-23 (Actual); Primary Completion 2020-02-28 (Actual); Study Completion 2020-02-28 (Actual)

PRIMARY OUTCOMES:
Changes in gaming-related positive emotional association biases (EAB) | baseline , the 1st day after training
  The gaming-related positive EAB will be assessed in a priming task. In the task, participants will be instructed to judge the emotional valence of positive or negative words following gaming pictures or healthy-activity pictures. Gaming-related positive EAB will be calculated by determining differences in reaction times (RTs; RTs (negative-word) minus RTs (positive-word)) in response to words following gaming pictures
Changes in gaming-related compulsive thoughts | baseline, the 1st week after training, the 2nd week after training, the 3rd week after training, the 4th week after training, the 6th week after training, the 8th week after training
  the scores of gaming-related compulsive thoughts will be assessed with the Yale-Brown Obsessive-Compulsive Scale modified for internet gaming disorder. The range of the score concerning gaming-related compulsive thoughts of this scale is from 0 to 20. Higher scores means more gaming-related compulsive thoughts.
Changes in gaming-related compulsive behaviors | baseline, the 1st week after training, the 2nd week after training, the 3rd week after training, the 4th week after training, the 6th week after training, the 8th week after training
  the scores of gaming-related compulsive behaviors will be assessed with the Yale-Brown Obsessive-Compulsive Scale modified for internet gaming disorder. The range of the score concerning gaming-related compulsive behaviors of this scale is from 0 to 20. Higher scores means more gaming-related compulsive behaviors.

SECONDARY OUTCOMES:
Changes in positive healthy-activity-related EAB | baseline and the 1st day after training
  The healthy-activity-related positive EAB will be assessed in a priming task. In the task, participants will be instructed to judge the emotional valence of positive or negative words following gaming pictures or healthy-activity pictures. Healthy-activity-related positive EAB will be calculated by determining differences in reaction times (RTs; RTs (negative-word) minus RTs (positive-word)) in response to words following healthy-activity pictures
Changes in IGD severity | baseline, the 4th week after training, the 8th week after training
  The scores of IGD severity will be assessed with the internet addiction test for internet gaming disorder. The range of the score of this scale is from 20 to 100. Higher scores means severer internet gaming disorder.
Changes in weekly gaming time | baseline, the 1st week after training, the 2nd week after training, the 3rd week after training, the 4th week after training, the 6th week after training, the 8th week after training
  weekly gaming time will be assessed by instructing participants to report weekly gaming hour in a questionaire
Changes in craving | baseline , the 1st day after training
  In the regulation-of-craving task, participants will report gaming-related craving during look condition, and during regulation condition using cognitive reappraisal，respectively. Craving will be assessed using a Visual Analog Scale (from 1 = 'not at all' to 9 = 'very high')

CONTACTS AND LOCATIONS:
Overall Officials: Jintao Zhang, phD, Principal Investigator — Beijing Normal University
Locations (1):
- State Key Laboratory of Cognitive Neuroscience and Learning, Beijing Normal University, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Yes
we will share individual participant data when required
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 1 year after the publication of related paper , for 3 years
Access Criteria: By contacting the principal investigator. Email : zhangjintao@bnu.edu.cn

REFERENCES:
- [Background] Snagowski J, Wegmann E, Pekal J, Laier C, Brand M. Implicit associations in cybersex addiction: Adaption of an Implicit Association Test with pornographic pictures. Addict Behav. 2015 Oct;49:7-12. doi: 10.1016/j.addbeh.2015.05.009. Epub 2015 May 16. PMID 26026385
- [Derived] Wu L, Xu J, Song K, Zhu L, Zhou N, Xu L, Liu G, Wang Z, Wang R, Qin S, Fang X, Zhang J, Potenza MN. Emotional bias modification weakens game-related compulsivity and reshapes frontostriatal pathways. Brain. 2022 Dec 19;145(12):4210-4221. doi: 10.1093/brain/awac267. PMID 35861265